CLINICAL TRIAL: NCT00447083
Title: A Pilot Study of the Effect of Ultraviolet Light on Pain in Persons With Fibromyalgia Syndrome
Brief Title: Benefits of Tanning in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: II-CDR-Fibromyalgia
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-10

CONDITIONS: Fibromyalgia Syndrome
Keywords: Tanning; Musculoskeletal; Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- UVB First (Experimental): Subjects with fibromyalgia will undergo 6 tanning sessions (3/week x 2 weeks) at which they will be exposed in tanning beds with UV. The dose of UV (time of exposure) will be progressively increased from 3 minutes to 9 minutes over the 6 visits to acclimate subjects to UV light. Before and after every tanning session the subject will complete the pain questionnaire. Subjects in this group will be randomized to receive UVB tanning bed treatment first, then switch to the non-UVB treatment.
  Interventions: Device: UVB; Procedure: Non-UVB
- Non-UVB First (Placebo Comparator): Subjects with fibromyalgia will undergo 6 tanning sessions (3/week x 2 weeks) at which they will be exposed in tanning beds with non-UV bulbs. The time of exposure will be progressively increased from 3 minutes to 9 minutes over the 6 visits to mirror UVB treatment. Before and after every tanning session the subject will complete the pain questionnaire. Subjects in this group will be randomized to receive non-UVB tanning bed treatment first, then switch to the UVB treatment.
  Interventions: Device: UVB; Procedure: Non-UVB
- UVB (Experimental): The subjects who complete the acclimation phase of the study will then be randomized to 3 times/week treatments for 6 weeks with a fixed dose (10 min) of UVB.
  Interventions: Device: UVB
- Non-UVB (Placebo Comparator): The subjects who complete the acclimation phase of the study will then be randomized to 3 times/week treatments for 6 weeks with a fixed dose (10 min) of non-UVB exposure
  Interventions: Procedure: Non-UVB

INTERVENTIONS:
Device: UVB — UVB exposure by a tanning bed
  Other Names: Ultraviolet Light
  Arms: Non-UVB First; UVB; UVB First
Procedure: Non-UVB — Non-UVB exposure by a tanning bed
  Arms: Non-UVB; Non-UVB First; UVB First

SUMMARY:
* To establish whether ultraviolet light exposure acutely reduces perceptions of pain in patients with fibromyalgia.
* To establish whether a series of UV light exposures has a cumulative effect on fibromyalgia pain.

DETAILED DESCRIPTION:
Fibromyalgia is a common chronic disorder characterized by widespread pain and fatigue. It occurs primarily in women, especially women of childbearing age. The effectiveness of treatment for this disorder is limited, and alternative medical treatments are commonly used.

Ultraviolet (UV) light exposure gives a sense of relaxation. It is unknown whether UV exposure has any effect on pain, particularly in patients with fibromyalgia. Through studies performed with RO3 funding from the National Institute of Drug Abuse (NIDA), we demonstrated that in frequent tanners, appearance is less important than UV-induced relaxation in motivating tanning behavior. Moreover, we determined that UV light has reinforcing properties apart from any psychosocial benefits of having a tan. One subject in our study reported low back pain relief from the UV exposure condition.

This is a two-year proposal that is the beginning of a long-term plan to assess whether indoor tanning ultraviolet light exposure has a therapeutic effect for patients with chronic pain. To this end, we will determine the effect of UV light on fibromyalgia pain in a controlled, double blind clinical trial of UV exposure. This approach is carefully designed to separate the effects of UV exposure on pain from potential confounds associated with the tanning procedure, including any perceived benefits of having a tan. The results of this study will increase our understanding of the specific influence of UV light on persistence in tanning behavior.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia patients who meet the fibromyalgia criteria, and who have been diagnosed with fibromyalgia by a board certified rheumatologist. The fibromyalgia criteria {as defined by the American College of Rheumatology (ACR)} require the patient to have: at least 3 months of widespread pain defined as: bilateral; above and below the waist, including axial skeletal pain; and pain to palpation with 4kg of pressure at a minimum of 11 out of 18 predefined tender points.
* Ideally, patients should not be taking medication for treatment of fibromyalgia, and they should not be taking psychoactive medications on an as needed basis for treatment of fibromyalgia. However, if patients are taking psychoactive or other medications for the treatment of fibromyalgia, then they should be on a stable dose, defined as no change in dosage in the 4 weeks prior to study enrollment.
* Patients must agree to not partake in tanning bed UV exposure during the study.

Exclusion Criteria:

* Fitzpatrick skin type 1 ("never tan, always burn")
* Past or present skin cancer
* Current use of photosensitizing drugs (current use of photosensitizing drugs will be evaluated via a patient questionnaire at time of patient enrollment - see Appendix 1),, psychoactive medications (not a stable dose, defined as no change in dosage in the 4 weeks prior to study enrollment), or illicit drugs
* Pregnant, planning to become pregnant, or breast feeding
* Significant visual discrimination of UV versus non-UV conditions
* Greater than 6 indoor tanning sessions over the past year
* Concurrent photosensitive disease, positive antinuclear antibody test, positive anti-Smith antibody test, or positive anti-dsDNA test.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2005-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Feldman, M.D., Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - UVB First: Subjects with fibromyalgia will undergo 6 tanning sessions (3/week x 2 weeks) at which they will be exposed in tanning beds with UV. The dose of UV (time of exposure) will be progressively increased from 3 minutes to 9 minutes over the 6 visits to acclimate subjects to UV light. Before and after every tanning session the subject will complete the pain questionnaire. Subjects in this group will be randomized to receive UVB tanning bed treatment first, then switch to the non-UVB treatment.
  UVB: UVB exposure by a tanning bed
- Phase I - Non-UVB First: Subjects with fibromyalgia will undergo 6 tanning sessions (3/week x 2 weeks) at which they will be exposed in tanning beds with non-UV bulbs. The time of exposure will be progressively increased from 3 minutes to 9 minutes over the 6 visits to mirror UVB treatment. Before and after every tanning session the subject will complete the pain questionnaire. Subjects in this group will be randomized to receive non-UVB tanning bed treatment first, then switch to the UVB treatment.
  UVB: UVB exposure by a tanning bed
- Phase II - UVB Exposure: Part of the subjects who complete the acclimation phase of the study ( Phase I) will then be randomized to 3 times/week treatments for 6 weeks with a fixed dose (10 min) of UVB.
- Phase II -Non-UVB: Part of the subjects who complete the acclimation phase of the study ( Phase I) will then be randomized to 3 times/week treatments for 6 weeks with a fixed dose (10 min) of non-UVB exposure in Phase II.
Period: Phase I
Arm/Group | Phase I - UVB First | Phase I - Non-UVB First | Phase II - UVB Exposure | Phase II -Non-UVB
Started | 10 | 9 | 0 | 0
Completed | 10 (2 participants did not acclimate to phase II) | 9 (1 participant did not acclimate to phase II) | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I - UVB First | Phase I - Non-UVB First | Phase II - UVB Exposure | Phase II -Non-UVB
Started | 0 (Participants in this group will then be randomized to a phase 2 group in phase2) | 0 (Participants in this group will then be randomized to a phase 2 group in phase2) | 8 (Only 8 participants qualified from the end of phase 1) | 8 (Only 8 participants qualified from the end of phase 1)
Completed | 0 | 0 | 7 | 7
Not Completed | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UVB First | Non-UVB First | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief Success Rates (Phase I)
Description: Percentage of exposures that showed pain relief (2 point improvement in Likert scale) in the 11 point Likert scale.
Time Frame: 2 weeks
Measure: Number; unit: percentage of exposures with relief
Groups:
- UVB Exposure: Subjects with fibromyalgia will undergo 6 tanning sessions (3/week x 2 weeks) at which they will be exposed in tanning beds with UV. The dose of UV (time of exposure) will be progressively increased from 3 minutes to 9 minutes over the 6 visits to acclimate subjects to UV light. Before and after every tanning session the subject will complete the pain questionnaire. Subjects in this group received UVB tanning bed treatment.
  UVB: UVB exposure by a tanning bed
- Non-UVB Exposure: Subjects with fibromyalgia will undergo 6 tanning sessions (3/week x 2 weeks) at which they will be exposed in tanning beds with non-UV bulbs. The time of exposure will be progressively increased from 3 minutes to 9 minutes over the 6 visits to mirror UVB treatment. Before and after every tanning session the subject will complete the pain questionnaire. Subjects in this group received non-UVB tanning bed treatment.
  UVB: UVB exposure by a tanning bed
Arm/Group | UVB Exposure | Non-UVB Exposure
Number analyzed (Participants) | 19 | 19
percentage of exposures with relief | 33 | 16

2. Primary Outcome: Pain Score- Likert Scale(Phase II)
Description: Pain will be assessed on an 11-point pain scale where 0=no pain and 10=worst possible pain. A 30% improvement in reported pain will be considered a treatment "success.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- UVB Exposure: The subjects who complete the acclimation phase of the study will then be randomized to 3 times/week treatments for 6 weeks with a fixed dose (10 min) of UVB.
Arm/Group | UVB Exposure | Non-UVB
Number analyzed (Participants) | 7 | 7
score on a scale | 4.55 (0.29) | 4.95 (0.24)

3. Secondary Outcome: Post-treatment Pain Scores- Likert Scale (Phase I)
Description: As a secondary outcome, the post-treatment pain scores between the UV and non-UV exposures given on the first day the dose is given will be compared. Pain will be assessed on an 11-point pain Likert scale where 0=no pain and 10=worst possible pain
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UVB Exposure | Non-UVB Exposure
Number analyzed (Participants) | 19 | 19
score on a scale | 4.89 (2.56) | 5.21 (2.64)

4. Secondary Outcome: Pain Scores of the UV and Non-UV Exposure (Phase II)
Description: The pain scores were assessed using a Likert Scale. Pain will be assessed on an 11-point pain Likert scale where 0=no pain and 10=worst possible pain.
Time Frame: 4 weeks post-treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | UVB Exposure | Non-UVB
Number analyzed (Participants) | 7 | 7
score on a scale | 4.65 (.56) | 5.54 (.32)
Statistical Analysis 1: Comparison: UVB Exposure vs Non-UVB; Test type: Other; p = .1811, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | UVB Exposure | Non-UVB
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes